CLINICAL TRIAL: NCT04334460
Title: Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Antiviral Activity of BLD-2660 in Hospitalized Subjects With Recently Diagnosed COVID-19 Compared to Standard of Care Treatment
Brief Title: Safety and Antiviral Activity of BLD-2660 in COVID-19 Hospitalized Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Blade Therapeutics (Industry)
Collaborators: Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-2660-204
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-02

CONDITIONS: Sars-CoV-2; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (BLD-2660) Group (Active Comparator)
  Interventions: Drug: BLD-2660
- Placebo Group (Placebo Comparator)
  Interventions: Drug: BLD-2660

INTERVENTIONS:
Drug: BLD-2660 — BLD-2660 is a novel, synthetic, orally active, small molecule inhibitor of calpain (CAPN) 1, 2, and 9.

SUMMARY:
BLD-2660 is a novel, synthetic, orally active, small molecule inhibitor of calpain (CAPN) 1, 2, and 9 that is selective over the cathepsins as well as other protease families, displays good metabolic stability and permeability, oral bioavailability and low cytochrome P450 (CYP) inhibition. It is under development for the treatment of coronavirus disease-19 (COVID-19) resulting from infection with Severe Acute Respiratory Syndrome Coronavirus 2 (SARSCoV2), where there is significant unmet medical need.

DETAILED DESCRIPTION:
Interleukin 6 (IL-6), a proinflammatory cytokine, is a key driver of a cytokine storm that plays a significant role in clinical complications and acute lung injury. Emerging data indicate that serum levels of IL-6 are elevated in COVID-19 patients and are predictive of respiratory failure and mortality. IL-6 has been shown to contribute to lung damage during SARS-CoV infection and the virus itself is capable of directly inducing its expression. Suppression of pro-inflammatory IL-6 have been shown to have a therapeutic effect in many inflammatory diseases, including viral infections.

In a mouse model of lung injury employing bleomycin, BLD-2660, at therapeutic doses of 30 and 100 mg/kg twice per day (BID), reduced IL-6 levels in bronchoalveolar lavage (BAL) fluid. BLD-2660 also attenuated fibrosis damage as measured by significant reductions in the alpha smooth muscle actin and collagen 1 in lung tissue. BLD-2660 also demonstrated target engagement by inhibiting cleavage of one of its substrates, spectrin, in bronchoalveolar cells.

BLD-2660 was also evaluated in a mouse model of NASH fibrosis, demonstrating an anti-fibrotic effect. A significant decrease in IL-6 transcription was also observed. This suggests that the effect of BLD-2660 on IL-6 is independent of the injury, or the affected organ.

It has been shown that the receptor for SARS-CoV-1 and -2 entry into the cell is angiotensin-converting enzyme 2 (ACE-2). ACE-2 and the dimeric calpains (data on file) are co-expressed in respiratory epithelial cells, the site of both viral entry and predominant early lung injury in COVID-19. Inhibition of dimeric calpain activity has not been associated with impairment of normal immune function. The safety and tolerability of BLD-2660 has been demonstrated in the recently completed Phase 1 single ascending dose (SAD)/multiple ascending dose (MAD) B-2660-101 study.

As BLD-2660 has been demonstrated to (1) reduce tissue IL-6 levels and (2) attenuate lung fibrosis damage, it could therefore, potentially reduce the nonproductive IL-6 mediated host-response to infection, which contribute to morbidity and mortality in COVID-19. In addition, data suggest that survivors of SARS-CoV-2 infection are at risk for chronic impairment of pulmonary function, likely attributable to pulmonary fibrosis secondary to lung injury and inflammation. Although there is not yet available data documenting numbers of patients infected with SARS CoV2 pneumonia who progress to pulmonary fibrosis, epidemiology, viral immunology, and current clinical evidence support that pulmonary fibrosis may become one of the serious long-term complications of survivors of COVID-19 related pneumonia.

Thus, BLD-2660 could not only potentially downregulate the nonproductive host-response to infection, which contributes to morbidity and mortality in COVID-19 but also could reduce potential long-term fibrosis and loss of pulmonary function resulting from SARS-CoV pneumonia. This study will evaluate BLD-2660 as an add-on therapy to standard of care (SOC) in hospitalized subjects with recent diagnosis of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

At least 18 years of age at the time of signing the ICF.

Hospitalized for COVID-19.

Diagnosed with COVID-19 as defined by having at least 2 of the following signs or symptoms within the past 2 days:

* Fever defined as a body temperature of ≥ 38.0 °C oral, or ≥ 38.3 °C rectal, ≥37.7 °C forehead or ≥38.7°C aural (axillary temperatures are not allowable);
* Cough;
* Fatigue;
* Shortness of breath.

Radiographic evidence (chest x-ray or CT scan) of one the following:

* Ground-glass opacities, or
* Local or bilateral patchy infiltrates, or
* Interstitial pulmonary infiltrates.

Oxygen requirements:

* SpO2 ≤ 94% on ambient air OR
* Requires supplemental oxygen administration by nasal cannula, simple face mask, or other similar oxygen delivery device.

Male and/or female subjects.

- Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

All subjects (male or female) who are of childbearing potential must agree to use highly effective contraception during the study. Female subjects and male partners of female subjects must continue to use highly effective contraception for 30 days after the last dose of study drug. Female subjects should not donate oocytes during this time. Male subjects and female partners of male subjects must continue to use highly effective contraception for 90 days. Male subjects must agree not to donate sperm during this time.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Note: Ethinyl estradiol is the primary estrogen used in hormonal contraceptives. The progestin component consists of norethindrone, levonorgestrel, norgestrel, norethindrone acetate, ethynodiol diacetate, norgestimate, desogestrel, and drospirenone. As BLD-2660 is a weak CYP3A4 inducer, exposure to both the estrogen and progestin components in hormonal contraceptives may be decreased, resulting in an increased risk of pregnancy. As such, it is recommended that subjects who are on hormonal contraceptives for birth control should use an alternate means of contraception (condoms, diaphragms, intrauterine device (IUD), other barrier methods, sexual abstinence, etc.) during participation in the study.

Women of childbearing potential must have a negative serum pregnancy test at Screening within 72 hours prior to first administration of study drug.

Women not of childbearing potential must be postmenopausal (defined as cessation of regular menstrual periods for at least 1 year

Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol

Exclusion Criteria:

Active bacterial pneumonia infection

Known active tuberculosis (TB).

History of Child-Pugh B or C cirrhosis.

History of ischemic heart disease or myocardial infarction or acute coronary syndrome.

Subjects requiring supplemental oxygen ≥0.75 FiO2.

It is not in the best interest of the subjects to participate, in the opinion of the treating Investigator.

Female subjects who are pregnant or breastfeeding or expecting to conceive within the projected duration of the study, starting with the screening visit through 90 days after the last dose of study drug.

The following laboratory parameters are excluded:

* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 x upper limit of normal (ULN);
* Creatinine clearance < 50 mL/min.

Requiring, or expected to require mechanical ventilation at screening.

Treatment with chloroquine or hydroxychloroquine at study entry.

Treatment with anti-IL 6, anti-IL-6 receptor antagonists, or with Janus kinase inhibitors (JAKi) in the past 30 days or plans to receive during the study period.

Participation in any other clinical study of an experimental drug treatment for COVID-19 within 6 half-lives of the experimental treatment.

Note: Subjects participating in an observational study are an exception to this criterion and may qualify for the study with Sponsor approval.

Note: Subjects who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Unable to swallow solid oral medication or known malabsorption disorder.
* Subjects who have allergy to BLD-2660 or inactive components of BLD-2660.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (26):
  - Blade Research Site, Irvine, California
  - Blade Research Site, Los Angeles, California
  - Blade Reseach Site, San Jose, California
  - Blade Research Site, Washington D.C., District of Columbia
  - Blade Research Site, Brandon, Florida
  - Blade Research Site, Ft. Pierce, Florida
  - Blade Research Site, Panama City, Florida
  - Blade Research Site, Tampa, Florida
  - Blade Research Site, Idaho Falls, Idaho
  - Blade Research Site, Peoria, Illinois
  - Blade Research Site, Ames, Iowa
  - Blade Research Site, Lexington, Kentucky
  - Blade Research Site, Louisville, Kentucky
  - Blade Research Site, Baltimore, Maryland
  - Blade Research Site, Detroit, Michigan
  - Blade Research Site, Farmington Hills, Michigan
  - Blade Research Site, Omaha, Nebraska
  - Blade Research Site, Ridgewood, New Jersey
  - Blade Research Site, Charleston, North Carolina
  - Blade Research Site, Durham, North Carolina
  - Blade Research Site, Fayetteville, North Carolina
  - Blade Research Site, Philadelphia, Pennsylvania
  - Blade Research Site, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Blade Research Site, Dallas, Texas
  - Blade Research Site, Spokane, Washington
- Brazil (8):
  - Blade Research Site, Campinas, São Paulo
  - Blade Research Site, Bahia
  - Blade Research Site, Belo Horizonte
  - Blade Research Site, Botucatu
  - Blade Research Site, Porto Velho
  - Blade Research Site, Ribeirão Preto
  - Blade Research Site, São José do Rio Preto
  - Blade Research Site, Vitória

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Group: BLD-2660: BLD-2660 is a novel, synthetic, orally active, small molecule inhibitor of calpain (CAPN) 1, 2, and 9.
- Placebo Group: Placebo: Placebo-to-Match BLD-2660
Period: Full Enrollment
Arm/Group | Active Group | Placebo Group
Started | 81 | 39
Completed | 81 | 39
Not Completed | 0 | 0
Period: Full Analysis Set (FAS)
Arm/Group | Active Group | Placebo Group
Started | 81 | 39
Completed | 77 | 38
Not Completed | 4 | 1
Not completed — Patients did not receive any study drug & are therefore excluded from the FAS. | 4 | 1
Period: Safety Analysis Population
Arm/Group | Active Group | Placebo Group
Started | 81 | 39
Completed | 77 | 38
Not Completed | 4 | 1
Not completed — Patients did not receive any study drug & are therefore excluded from the Safety analysis set. | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: Placebo to Match (PTM) the active BLD-2660
- Total: Total of all reporting groups
Arm/Group | Active Group | Placebo Group | Total
Number analyzed (Participants) | 81 | 39 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (12.97) | 54.2 (13.95) | 52.2 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 13 | 55
  Male | 39 | 26 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 19 | 64
  Not Hispanic or Latino | 35 | 19 | 54
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 13 | 11 | 24
  White | 60 | 20 | 80
  More than one race | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 19 | 59
  Brazil | 41 | 20 | 61
APACHE II Score [Mean (Standard Deviation); unit: units on a scale] — The Acute Physiology and Chronic Health Evaluation Two Score (APACHE II) is a severity score and mortality estimation tool for predicting mortality. The APACHE II score ranges from 0 to 71 and is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death. For example, a score of 25 represents a predicted mortality of 50% and a score of over 35 represents a predicted mortality of 80%. Population: The reason is due to missing data.
  units on a scale
    number analyzed (Participants) | 71 | 31 | 102
    (all) | 6.5 (5.41) | 6.5 (4.84) | 6.5 (5.22)
6-Point Ordinal Scale [Count of Participants; unit: Participants] — Population: The reason is due to missing data.
  Participants
    number analyzed (Participants) | 77 | 38 | 115
    1 - Not hospitalized | 0 | 0 | 0
    2 - Hospitalized, not requiring supplemental oxygen | 6 | 1 | 7
    3 - Hospitalized, requiring supplemental oxygen | 60 | 25 | 85
    4 - Hospitalized, on non-invasive ventilation or high flow oxygen device | 6 | 7 | 13
    5 - Hospitalized, on invasive mechanical ventilation or ECMO | 0 | 0 | 0
    6 - Death | 0 | 0 | 0
    7 - Missing | 5 | 5 | 10
SpO2/FiO2 Ratio [Mean (Standard Deviation); unit: Ratio] — Population: The reason is due to missing data.
  Ratio
    number analyzed (Participants) | 72 | 37 | 109
    (all) | 299.2 (61.89) | 290.8 (72.34) | 296.3 (65.41)
SARS-Cov-2 PCR Viral Load (copies/mL) [Mean (Standard Deviation); unit: copies/mL] — Population: The reason is due to missing data.
  copies/mL
    number analyzed (Participants) | 71 | 34 | 105
    (all) | 5703533.3 (30719776.01) | 553963.0 (2177374.66) | 4036053.4 (25348615.41)
IL-6 (ng/mL) [Mean (Standard Deviation); unit: ng/mL] — Population: The reason is due to missing data.
  ng/mL
    number analyzed (Participants) | 70 | 35 | 105
    (all) | 12.9 (27.60) | 11.3 (13.10) | 12.4 (23.71)
D-Dimer (ug/mL) [Mean (Standard Deviation); unit: ug/mL] — Population: The reason is due to missing data.
  ug/mL
    number analyzed (Participants) | 64 | 33 | 97
    (all) | 0.8 (0.70) | 0.8 (0.62) | 0.8 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery
Description: To evaluate time to recovery as defined by no longer requiring oxygen support or hospital discharge, whichever occurs first.
Time Frame: Course of study; 28 days
Population: FAS Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 77 | 38
days | 5 [3.00 to 6.00] | 4.5 [4.00 to 6.00]

2. Primary Outcome: Change in Oxygenation
Description: To evaluate change in oxygenation in hospitalized adults with COVID-19 treated with BLD-2660. Measured by change from baseline to Day 10 or hospital discharge, if sooner, in the ratio of peripheral hemoglobin oxygen saturation to fraction of inspired oxygen (SpO2/FiO2)
Time Frame: 10 days
Population: FAS Set
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 77 | 38
Ratio | 33.8 (17.10) | 66.8 (25.58)

3. Secondary Outcome: Safety & Tolerability: Incidence of TEAEs and Serious Adverse Events (SAEs)
Description: To evaluate the safety and tolerability of BLD-2660 in the same population. Measured by incidence of TEAEs and serious adverse events (SAEs)
Time Frame: Course of study; 28 days
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 77 | 38
Participants
  Number of Subjects with >=1 TEAE | 42 | 23
  Number of Subjects with >=1 Treatment-Related TEAE | 10 | 6
  Number of Subjects with >=1 TEAE with Grade 3 or higher | 12 | 9
  Number of Subjects with >=1 TE SAE | 9 | 9
  Number of Subjects with >=1 Treatment-Related SAE | 0 | 1
  Number of Subjects with >=1 TEAE leading to discontinuation of study drug | 2 | 5
  Number of fatal AEs | 2 | 2

4. Other Pre Specified Outcome: Time to Discharge Readiness
Description: Measured by time to discharge readiness
Time Frame: Course of study; 28 days
Population: FAS Set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 77 | 38
Days | 7.0 [6.00 to 11.00] | 8.0 [5.00 to 22.00]

5. Other Pre Specified Outcome: Proportion of Subjects Discharged During Study
Description: Measured by proportion of subjects ready to be discharged from the hospital during the 28-day study period following enrollment.
Time Frame: Course of study; 28 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Time to Resolution of Fever
Description: Measured by time to resolution of fever below entry criteria for 24 hours in subjects with fever at baseline
Time Frame: Course of study; 28 days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Duration of Remdesivir Use
Description: Measured by duration (in days) of remdesivir use in subjects starting remdesivir within 24 hours of first dose of BLD-2660
Time Frame: Course of study; 28 days
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Clinical Status
Description: Measured by change from baseline to Days 10, 14, 21 and 28 in clinical status outcome using a 6-point ordinal scale
Time Frame: Course of study; 28 days
Population: FAS Set
Measure: Count of Participants; unit: Participants
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 77 | 38
Participants
  Day 10/EOT: 1 - Not hospitalized | 4 | 0
  Day 10/EOT: 2 - Hospitalized, not requiring supplemental oxygen | 44 | 23
  Day 10/EOT: 3 - Hospitalized, requiring supplemental oxygen | 20 | 8
  Day 10/EOT: 4 - Hospitalized, on non-invasive ventilation or high flow oxygen device | 3 | 3
  Day 10/EOT: 5 - Hospitalized, on invasive mechanical ventilation or ECMO | 5 | 2
  Day 10/EOT: 6 - Death | 0 | 0
  Day 10/EOT: 7 - Missing | 1 | 2
  Day 14 (Follow-Up): 1 - Not hospitalized | 56 | 21
  Day 14 (Follow-Up): 2 - Hospitalized, not requiring supplemental oxygen | 5 | 2
  Day 14 (Follow-Up): 3 - Hospitalized, requiring supplemental oxygen | 1 | 1
  Day 14 (Follow-Up): 4 - Hospitalized, on non-invasive ventilation or high flow oxygen device | 3 | 1
  Day 14 (Follow-Up): 5 - Hospitalized, on invasive mechanical ventilation or ECMO | 3 | 2
  Day 14 (Follow-Up): 6 - Death | 0 | 0
  Day 14 (Follow-Up): 7 - Missing | 9 | 11
  Day 21 (Follow-Up): 1 - Not hospitalized | 54 | 20
  Day 21 (Follow-Up): 2 - Hospitalized, not requiring supplemental oxygen | 2 | 1
  Day 21 (Follow-Up): 3 - Hospitalized, requiring supplemental oxygen | 1 | 1
  Day 21 (Follow-Up): 4 - Hospitalized, on non-invasive ventilation or high flow oxygen device | 0 | 0
  Day 21 (Follow-Up): 5 - Hospitalized, on invasive mechanical ventilation or ECMO | 3 | 1
  Day 21 (Follow-Up): 6 - Death | 0 | 0
  Day 21 (Follow-Up): 7 - Missing | 17 | 15
  Day 28: 1 - Not hospitalized | 63 | 24
  Day 28: 2 - Hospitalized, not requiring supplemental oxygen | 0 | 1
  Day 28: 3 - Hospitalized, requiring supplemental oxygen | 1 | 0
  Day 28: 4 - Hospitalized, on non-invasive ventilation or high flow oxygen device | 0 | 0
  Day 28: 5 - Hospitalized, on invasive mechanical ventilation or ECMO | 3 | 1
  Day 28: 6 - Death | 0 | 0
  Day 28: 7 - Missing | 10 | 12

9. Other Pre Specified Outcome: Percentage of Subjects in Each Category of the 6-point Ordinal Scale
Description: Measured by percentage of subjects reporting each 6-point ordinal scale of the clinical status outcome assessment.
Time Frame: Course of study; 28 days
Population: FAS Set
Measure: Count of Participants; unit: Participants
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 77 | 38
Participants
  Day 10 (EOT) | 76 | 36
  Day 14 (Follow-Up) | 68 | 27
  Day 21 (Follow-Up) | 60 | 23
  Day 28 | 67 | 26

10. Other Pre Specified Outcome: Change in IL-6
Description: Measured by change from baseline to Days 10, 14, 21 and 28 in IL-6 in ng/mL measured by analytical assay
Time Frame: Course of study; 28 days
Population: FAS Set. Only participants in the FAS with data at the respective time point are summarized.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 77 | 38
ng/L
  Day 10: number analyzed (Participants) | 64 | 34
  Day 10 | 5.606 (13.6212) | 4.592 (8.8388)
  Day 14: number analyzed (Participants) | 57 | 23
  Day 14 | 29.547 (196.4762) | 25.892 (82.0965)
  Day 21: number analyzed (Participants) | 49 | 18
  Day 21 | 3.361 (6.6323) | 1.981 (1.9770)
  Day 28: number analyzed (Participants) | 49 | 20
  Day 28 | 6.639 (28.6087) | 2.649 (4.0756)

11. Other Pre Specified Outcome: Change in D-dimer
Description: Measured by change from baseline to Days 10, 14, 21 and 28 in D-dimer in ng/mL measured by analytical assay
Time Frame: Course of study; 28 days
Population: FAS Set
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 77 | 38
ug/mL
  Day 10: number analyzed (Participants) | 57 | 29
  Day 10 | 0.51 [0.404 to 0.646] | 0.67 [0.488 to 0.926]
  Day 14: number analyzed (Participants) | 58 | 23
  Day 14 | 0.54 [0.431 to 0.677] | 0.57 [0.409 to 0.805]
  Day 21: number analyzed (Participants) | 53 | 23
  Day 21 | 0.50 [0.391 to 0.6529] | 0.56 [0.398 to 0.783]
  Day 28: number analyzed (Participants) | 60 | 24
  Day 28 | 0.57 [0.456 to 0.719] | 0.41 [0.295 to 0.574]

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Active Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 2/77 | 2/38
Serious Adverse Events (participants affected / at risk) | 9/77 | 9/38
Other Adverse Events (participants affected / at risk) | 42/77 | 23/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Group (N=77) | Placebo Group (N=38)
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Acinetobacter bacteraemia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Group (N=77) | Placebo Group (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Vessel puncture site bruise (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Fungal infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract candidiasis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 1
Fibrin D dimer increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 3
Migraine (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 2
Myasthenia gravis (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT04334460/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT04334460/SAP_001.pdf